CLINICAL TRIAL: NCT07022717
Title: A Universal Primary Care Based Pilot Intervention to Reduce Youth Overdose Risk
Brief Title: A Universal Primary Care Based Intervention to Reduce Youth Overdose Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-45731; R61DA062217 (NIH)
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Overdose
Keywords: Brief overdose prevention; Naloxone; Youth patients; Health care providers; Primary care
MeSH Terms: conditions — Drug Overdose | interventions — Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Providers randomized into this arm will complete a 45-minute intervention training. The training will occur either in person or via Zoom teleconference and include overdose prevention education, the pilot brief overdose prevention education intervention, intervention practice, and how to complete the fidelity checklist to be completed at the end of each visit.
  Interventions: Behavioral: Brief youth overdose prevention education; Other: Information about Naloxone
- Control group (Active Comparator): Providers randomized into this arm will deliver usual care to the youth patients.
  Interventions: Other: Usual standard of care

INTERVENTIONS:
Behavioral: Brief youth overdose prevention education — Providers in the intervention group will inform youth participants about: the risk factors for overdose, how to stay safe and prevent overdose, how to recognize an overdose, and how to respond to an overdose.
  Arms: Intervention group
Other: Information about Naloxone — Providers in the intervention group will inform youth participants how to use naloxone and offered a kit to take home.
  Other Names: Narcan
  Arms: Intervention group
Other: Usual standard of care — Participants will be provided usual care by providers in the control group.
  Arms: Control group

SUMMARY:
Adolescent (ages 10-19) overdose deaths are the third leading cause of pediatric death and continue to rise in the United States. Healthcare providers have regular and trusted relationships with youth and have experience in providing public health injury prevention counseling. Youth have different motivations for using drugs, and many who experience fatal overdose do not have a history of opioid use. Primary care pediatric providers regularly provide developmentally appropriate injury prevention counseling for leading causes of pediatric fatal and nonfatal injury such as drowning prevention and firearms safety. However, there are no recommended, evidence-based overdose prevention interventions for youth, including in health care settings, even though research supports pediatricians and youth-serving clinicians providing harm reduction strategies such as naloxone distribution and overdose education. Among adults, overdose prevention education reduces overdose, is cost-effective, and can be learned by laypersons. Content commonly includes awareness of fentanyl in the drug supply, risk reduction (e.g., not using alone, risks of polysubstance use), and how to recognize and respond to an overdose, including the use of naloxone.

This study is a pilot two-arm cluster randomized controlled trial (RCT) of a brief overdose prevention education intervention that will be developed in collaboration with the Community Advisory Board (CAB). The primary outcome of this study is to assess the feasibility and acceptability of the brief youth overdose prevention intervention as measured by provider feasibility and acceptability as well as youth acceptability.

ELIGIBILITY:
Inclusion Criteria for providers:

* Physicians and advance practice providers within Pediatric Primary Care and Family Medicine at Boston Medical Center (BMC)
* ≥ 2 clinic sessions per/week

Exclusion Criteria for providers:

* None

Inclusion criteria for youth:

* Ages 13-26
* Scheduled for a comprehensive physical exam with a provider who is participating in the trial
* English speaking

Exclusion criteria for youth:

* Caregivers of youth ages 13-17 unable to provide informed consent or are not English speaking
* Cognitive limitation or intellectual disability that in the opinion of their provider would not
* Any medical/psychiatric condition that causes acute distress and requires emergency evaluation
* Under legal custody of the Department of Children and Families (DCF)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the brief overdose prevention education intervention | 6 months
  Providers in the intervention arm will complete a checklist after all comprehensive physical exams with youth ages 13 to 26 years. The checklist will assess which components of the intervention the provider was able to deliver during the visit.
Provider acceptability of the brief overdose prevention education intervention | 6 months
  Providers in the intervention group will complete 8 questions based on the Theoretical Framework of Acceptability (TFA) acceptability questionnaire on a 5-point Likert scale. The measure will be collected post-intervention training and after all youth have received the intervention
Youth acceptability of the brief overdose prevention education intervention | 6 months
  Youth participants receiving care from providers in the interventions group will be asked after their comprehensive physical exam questions from an investigator developed questionnaire to rate their experience of the visit, receipt of the brief youth overdose prevention education intervention, importance, relevance, and comfort with the information.

SECONDARY OUTCOMES:
Youth perception of risk associated with fentanyl and other emerging drugs | Baseline, 2 weeks, 6-months
  A question assessing "Risk of taking medication you weren't prescribed" on a 3-point Likert scale adapted from the Monitoring the Future (MTF) survey
Youth awareness of strategies to reduce overdose risk | Baseline, 2 weeks, 6-months
  This outcome will be assessed by responses to an investigator developed questionnaire.
Youth's ability to recognize an overdose | Baseline, 2 weeks, 6-months
  This outcome will be assessed by responses to an investigator developed questionnaire.
Youth's ability to respond to an overdose | Baseline, 2 weeks, 6-months
  This outcome will be assessed by responses to an investigator developed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bagley, MD MSc, Principal Investigator — Boston Medical Center, Internal Medicine, Addiction Medicine; Amy Yule, MD, Principal Investigator — Boston Medical Center, Psychiatry
Locations (1):
- Boston Medical Center, Pediatric Primary Care & Family Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No